CLINICAL TRIAL: NCT01523496
Title: Vitamin D Supplementation and HIV-related Complications in Children and Young Adults
Brief Title: Vitamin D Supplementation in HIV Youth
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Grace McComsey, Professor of Pediatrics and Medicine, Chief Pediatric Infectious Diseases, Rheumatology and Global Health, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-11-06
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: HIV Infections
Keywords: HIV; Vitamin D Deficiency
MeSH Terms: conditions — HIV Infections; Vitamin D Deficiency | interventions — Calcifediol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV + Young Adults (Active Comparator): All will be HIV+ and receiving randomized dose of vitamin D control dose (low dose) or supplementation dose (vitamin D medium dose or vitamin D high dose)
  Interventions: Drug: Vitamin D control dose; Drug: Vitamin D supplementation-
- HIV - Controls (Active Comparator): HIV negative controls will be receiving randomized Vitamin D doses: control vitamin D dose (low dose) or vitamin D supplementation dose (vitamin D medium dose or vitamin D high dose)
  Interventions: Drug: Vitamin D control dose; Drug: Vitamin D supplementation-

INTERVENTIONS:
Drug: Vitamin D control dose — 18,000 IU per month
  Other Names: 25(OH)D3 low dose
Drug: Vitamin D supplementation- — 60,000 IU per month(medium dose) or 120,000 IU/month(high dose)
  Other Names: 25(OH)D3 medium dose or 25(OH)high dose

SUMMARY:
The purpose of this study is to determine the correct dose of Vitamin D to give to prevent HIV related complications.

DETAILED DESCRIPTION:
The purpose of the this study was to compare control dose of vitamin D (low dose of 600 IU/d) to supplementation dose (medium dose of 2000 IU/d or higher doses of vitamin D of 4000 IU/d) on HIV-related comorbidities including immune activation, inflammation, cardiovascular diseases, and metabolic complications in HIV-infected youth.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-25
* Documented HIV-1 infection
* On stable antiretroviral therapy for > 3 months
* Cumulative antiretroviral therapy of at least 6 months
* 25(OH)D level < 30 ng/ml at screening

Exclusion Criteria:

* > 400 IU daily regular vitamin D intake
* Parathyroid/calcium disorders
* Active malignancy
* Pregnancy/intent to become pregnant/breastfeeding
* Chronic infectious/inflammatory conditions
* Creatinine clearance < 50 ml/min
* Hemoglobin < 9.0 g/dL
* Aspartate aminotransferase and alanine aminotransferase > 2.5 upper limit of normal
* Diabetes requiring hypoglycemic agents
* Known coronary artery disease
* Inability to swallow pills

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 190 (Actual)
Dates: Start 2011-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, FIDSA, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - Emory Children's Center, Atlanta, Georgia
  - University Hospitals Case Medical Center, Cleveland, Ohio

REFERENCES:
- [Derived] Eckard AR, O'Riordan MA, Rosebush JC, Lee ST, Habib JG, Ruff JH, Labbato D, Daniels JE, Uribe-Leitz M, Tangpricha V, Chahroudi A, McComsey GA. Vitamin D supplementation decreases immune activation and exhaustion in HIV-1-infected youth. Antivir Ther. 2018;23(4):315-324. doi: 10.3851/IMP3199. PMID 28994661
- [Derived] Eckard AR, Rosebush JC, O'Riordan MA, Graves CC, Alexander A, Grover AK, Lee ST, Habib JG, Ruff JH, Chahroudi A, McComsey GA. Neurocognitive dysfunction in HIV-infected youth: investigating the relationship with immune activation. Antivir Ther. 2017;22(8):669-680. doi: 10.3851/IMP3157. PMID 28327462
- [Derived] Hileman CO, Overton ET, McComsey GA. Vitamin D and bone loss in HIV. Curr Opin HIV AIDS. 2016 May;11(3):277-84. doi: 10.1097/COH.0000000000000272. PMID 26890209

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV+ With Vit D Supplementation: HIV-infected adults who were supplemented with vit D ( medium dose: 60,000 IU per month or vitamin D high dose: 120,000 IU/month ) were combined into the supplementation group and compared to the standard control vitamin D dose
- HIV+ Young Adults With Vitamin D Control Dose: HIV+ receiving Vitamin D low dose: 18,000 IU per month
- HIV - With Vitamin D Supplementation: HIV-uninfected adults who were supplemented with vitamin D: a medium dose of 60,000 IU per month or a higher dose of 120,000 IU/month.
- HIV - With Vitamin D Control Dose: HIV uninfected controls receiving Vitamin D low dose: 18,000 IU per month
Period: Overall Study
Arm/Group | HIV+ With Vit D Supplementation | HIV+ Young Adults With Vitamin D Control Dose | HIV - With Vitamin D Supplementation | HIV - With Vitamin D Control Dose
Started | 66 (The supplementation group includes medium and high dose vitamin D supplementation) | 36 | 58 (The supplementation group includes medium and high dose vitamin D supplementation) | 30
Completed | 56 | 32 | 46 | 27
Not Completed | 10 | 4 | 12 | 3

BASELINE CHARACTERISTICS:
Population: A total of 190 subjects were enrolled, including 102 HIV-infected subjects: 66 on vitamin D supplementation dose, 36 on vitamin D control dose and 88 healthy controls: 58 on vitamin D supplementation dose, 30 on vitamin D control dose. By design, groups were well matched for age, sex and race.
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV+ With Vit D Supplementation | HIV+ Young Adults With Vitamin D Control Dose | HIV - With Vitamin D Supplementation | HIV - With Vitamin D Control Dose | Total
Number analyzed (Participants) | 66 | 36 | 58 | 30 | 190
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 20.9 [17.0 to 23.6] | 19.9 [15.9 to 21.6] | 19.6 [14.4 to 23.2] | 18.4 [14.4 to 22.2] | 19.9 [15.5 to 23.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 20 | 15 | 72
  Male | 44 | 21 | 38 | 15 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 57 | 34 | 47 | 29 | 167
  White | 9 | 2 | 11 | 1 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 36 | 58 | 30 | 190

OUTCOME MEASURES:

1. Primary Outcome: Changes in Serum 25(OH)D3 Levels
Description: Evaluate the dose-related efficacy of correction of Vitamin D deficiency for 25(OH)D3 levels in a group of HIV-infected children and young adults and a matched healthy control group in a randomized controlled study of different dosing regimens of oral Vitamin D supplementation: control dose (18,000 IU per month) or supplemented dose (medium 60,000IU per month or high dose 120,000IU/month )
Time Frame: 6 months
Population: HIV-infected on vitamin D control or supplementation dose and matched HIV-uninfected group on control or supplementation dose
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- HIV Positive on Vit D Control Dose: HIV+ receiving low vitamin D dose 18,000 IU per month
- HIV Positive on Vit D Supplementation Dose: HIV-infected young adults receiving a supplementation dose of vitamin D (either medium dose of 60,000 IU per month or a high dose of 120,000 IU/month)
- HIV Negative on Vitamin D Control Dose: HIV negative controls receiving Vitamin D low dose: 18,000 IU per month
- HIV Negative on Vitamin D Supplementation Dose: HIV negative controls receiving Vitamin D medium dose: 60,000 IU per month or vitamin D high dose: 120,000 IU/month
Arm/Group | HIV Positive on Vit D Control Dose | HIV Positive on Vit D Supplementation Dose | HIV Negative on Vitamin D Control Dose | HIV Negative on Vitamin D Supplementation Dose
Number analyzed (Participants) | 32 | 56 | 27 | 46
ng/mL | 11 [6 to 20] | 22 [14 to 32] | 7.5 [4 to 13] | 25 [15 to 35]

2. Secondary Outcome: Changes in Vitamin D Binding Protein (VDBP)
Description: Evaluate the dose-related efficacy of vitamin D binding Protein in levels in the blood in a group of HIV-infected children and young adults and a matched healthy control group in a randomized controlled study of different dosing regimens of oral vitamin D supplementation.
Time Frame: 6 months
Population: HIV-infected children and young adults and matched healthy control group. Results were not analyzed were captured comparing HIV+ young adults on control or supplementation vit D to HIV - controls
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- HIV + on Vitamin D Control Dose: HIV+ receiving vitamin D low dose: 18,000 IU per month
- HIV + on Vit D Supplementation Dose: HIV+ receiving Vitamin D supplementation (medium dose: 60,000 IU per month or higher dose: 120,000 IU/month)
- HIV Negative on Vit D Control Dose: HIV negative controls on Vitamin D low dose: 18,000 IU per month
- HIV Negative on Vit D Supplementation Dose: HIV negative controls on vitamin D supplementation: medium dose of 60,000 IU per month or higher dose of 120,000 IU/month
Arm/Group | HIV + on Vitamin D Control Dose | HIV + on Vit D Supplementation Dose | HIV Negative on Vit D Control Dose | HIV Negative on Vit D Supplementation Dose
Number analyzed (Participants) | 32 | 56 | 27 | 46
ng/mL | 3.9 [-17.9 to 12] | -8.9 [-41.3 to 13.3] | -11.3 [-202 to 5.4] | -11.7 [-183.6 to -2.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study duration, at baseline, 6 months, and 12 months.
Description: The same definitions are used. Systematic assessments of adverse events were done at each visit date by questionnaires, physical exam and vitamin D levels assessment by the study team. In case of adverse events they were reported to the principal investigator and then assessed in Data Safety and Monitory Board regular meetings.
Groups:
- HIV + on Vitamin D Control Dose: HIV+ receiving vitamin D control dose ( low dose: 18,000 IU per month)
- HIV+ on Vitamin D Supplementation Dose: HIV+ receiving vitamin D supplementation doses (medium dose of 60,000 IU per month or higher dose of 120,000 IU/month)
- HIV - on Vitamin D Control Dose: HIV negative patients receiving vitamin D control dose (low dose of 18,000 IU per month)
- HIV- on Vitamin D Supplementation Dose: HIV negative patients receiving vitamin D supplementation doses (medium dose of 60,000 IU per month or higher dose of 120,000 IU/month)
Arm/Group | HIV + on Vitamin D Control Dose | HIV+ on Vitamin D Supplementation Dose | HIV - on Vitamin D Control Dose | HIV- on Vitamin D Supplementation Dose
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/66 | 0/58 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/66 | 0/30 | 0/58
Other Adverse Events (participants affected / at risk) | 0/36 | 0/66 | 0/30 | 0/58

LIMITATIONS AND CAVEATS:
Limitations to this study include the lack of adherence measures to study drug such as pill counts and the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No